CLINICAL TRIAL: NCT02498626
Title: Are Venous Saturations From the Central Venous Line, Venous Side of the Heart Lung Machine Interchangeable or Not With Mixed Venous Saturation From the Pulmonary Artery in Children Undergoing Open Heart Surgery?
Brief Title: Mixed Venous Oxygen Saturation From Central Venous Line, Venous Side of Heart Lung Machine and the Pulmonary Artery
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine, Assiut University
Other Study IDs: IRB000087110
Record Dates: First submitted 2015-06-24; First posted 2015-07-15 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-02

CONDITIONS: Heart Defects, Congenital
Keywords: mixed venous saturation; open heart surgery; children
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- venous saturations: venous saturations from the central venous line, venous side of the heart lung machine and from the pulmonary artery
  Interventions: Other: venous saturations

INTERVENTIONS:
Other: venous saturations — Samples of venous saturations from the central venous line (CVP), from venous side of the heart lung machine and from the pulmonary artery were taken at 10 min after being on CPB and after correction of the cardiac defects.

SUMMARY:
This study was designed to examine if venous saturations from the central venous line and from the venous side of the heart lung machine are interchangeable or not with mixed venous saturation from the pulmonary artery in children undergoing open heart surgery for correction of various congenital heart defects.

DETAILED DESCRIPTION:
Forty children aged from 1-15 years undergoing correction for different congenital heart procedures with cardiopulmonary bypass [CPB] were included in this study. Simultaneous samples were taken from the central venous line, pulmonary artery, and from venous side of the heart lung machine. Samples were taken after 10 minutes on full CPB and at the end of surgery before end of CPB. Bland and Altman plots were used to study the agreement between venous saturations.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age from 1-15 years undergoing correction for congenital heart defects with cardiopulmonary bypass

Exclusion Criteria:

* Any chest renal or hepatic problems

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: cardiac surgery for children with congenital heart defects
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bland and Altman Analysis was used to plot the difference in mixed oxygen saturation | intraoperative
  The agreement between these samples from the central venous line, venous side of the heart lung machine and from the pulmonary artery were done using bland and Altman Analysis

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, MD, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt